CLINICAL TRIAL: NCT02984280
Title: Specific Respiratory Infections as Triggers of Acute Medical Events: Time Series Analysis Using LabBase and Hospital Episode Statistics
Brief Title: Specific Respiratory Infections as Triggers of Acute Medical Events
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/0440
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-11

CONDITIONS: Influenza, Human; Respiratory Syncytial Virus Infections; Parainfluenza; Rhinovirus; Adenovirus; Human Metapneumovirus Pneumonia; Cardiovascular Diseases
MeSH Terms: conditions — Influenza, Human; Respiratory Syncytial Virus Infections; Paramyxoviridae Infections; Adenoviridae Infections; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate whether there is a population-level association between circulating respiratory viruses and NHS hospital admissions for acute vascular events using data from national infection surveillance and Hospital Episode Statistics.

DETAILED DESCRIPTION:
We will conduct a time series study correlating anonymised population level data on all samples from NHS laboratories testing positive for six common respiratory viruses with admissions to NHS hospitals in England for a range of cardiac and vascular outcomes over the time period 01/01/2004 to 31/12/2014. This will involve generating Poisson regression models controlling for factors such as seasonal and long-term trends, environmental temperature and humidity.

This study is funded by an Academy of Medical Sciences Starter Grant for Clinical Lecturers.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with a record of an eligible outcome (ICD-10 coded hospitalisation for myocardial infarction or stroke) within the study period aged 45+ years
* Any individual with a record of an eligible exposure (laboratory-confirmed respiratory virus) within the study period at any age

Exclusion Criteria:

* Outcome events occurring in people aged <45 years

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population of England who have received NHS care during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 787000 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Acute myocardial infarction | 01/01/2004 to 31/12/2014
  ICD-10 coded
Stroke | 01/01/2004 to 31/12/2014
  ICD-10 coded

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte MJ Warren-Gash, MRCP PhD, Principal Investigator — UCL
Locations (1):
- University College London (UCL), London, United Kingdom

REFERENCES:
- [Derived] Blackburn R, Zhao H, Pebody R, Hayward A, Warren-Gash C. Laboratory-Confirmed Respiratory Infections as Predictors of Hospital Admission for Myocardial Infarction and Stroke: Time-Series Analysis of English Data for 2004-2015. Clin Infect Dis. 2018 Jun 18;67(1):8-17. doi: 10.1093/cid/cix1144. PMID 29324996